CLINICAL TRIAL: NCT02770443
Title: Withdrawal of Beta- Blockers and ACE Inhibitors After Left Ventricular Systolic Function Recovery in Patient With Dilated Cardiomyopathy: A Randomized Control Trial.
Brief Title: Withdrawal of Medication in Recovered DCM
Acronym: WrecEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed to recruitment early as endpoints were reached on several participants
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Nadia Giannetti, Chief, Division of Cardiology, Director of Heart Function Clinic, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-284-MUHC
Record Dates: First submitted 2016-04-29; First posted 2016-05-12 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Dilated Cardiomyopathy
Keywords: Recovered LVEF; DCM
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Adrenergic beta-Antagonists; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Withdrawal of beta blockers and ACE inhibitors
  Interventions: Drug: withdrawal
- control (Placebo Comparator): no withdrawal, standard of care
  Interventions: Drug: standard of CARE

INTERVENTIONS:
Drug: withdrawal — withdrawal of beta blocker and ACE inhibitors
  Other Names: withdrawal ACE and beta blockers; discontinuation of ACE and beta blockers
  Arms: Treatment
Drug: standard of CARE — STANDARD OF CARE, NO WITHDRAWAL OF MEDICAL THERAPY
  Arms: control

SUMMARY:
Randomized study of medication withdrawal in patients who have recovered LV function in Dilated Cardiomyopathy.

DETAILED DESCRIPTION:
Importance of the study:

There is a growing population of patients with dilated cardiomyopathy (DCM) who had recovered left ventricular (LV) systolic function on medical therapy. Recent studies have shown a favorable clinical course in patients with DCM1-4. The heart failure (HF) guidelines states that discontinuation of medical therapy in this group of patients may be considered based on expert opinion. The safety of withdrawal of medical therapy needs further studies.

Hypothesis:

In Patients with dilated cardiomyopathy (DCM) who had recovery of the LV systolic function to a normal EF >50%, medical therapy withdrawal is attainable without Clinical deterioration or recurrence of LV systolic dysfunction.

Objective

1. To study the withdrawal of guideline directed medical therapy, specifically beta-blockers and ACE/ARB, in patients with DCM after recovery of LV EF.
2. Correlate the sustained recovery in LVEF after medication discontinuation with specific genetic markers of recovery.

Method:

Study design:

It is a multi-center, non-blinded, randomized Control trial (pilot) comparing withdrawal of medical therapy in patients with recovered LVEF (recEF) compared to patients continuing medical therapy. Therapeutic changes will occur in a 2:1 randomization at the Royal Victoria Hospital, the Montreal General Hospital and the Jewish General Hospital. Patient would be recruited from a Heart Function Clinic or the echocardiography lab.

Procedures:

Patient Selection:

Patient selection will be conducted through chart review, ECHO lab, as well as the clinical visits. The DPS authorization will be requested.

Informed consent:

At time of enrolment the study's objective, procedures as well as the risks and benefits will be explained to the patient. A consent form will be provided to the patient. In addition, a wallet card and a medication discontinuations chart.

Randomization:

Randomization will be conducted in 2:1 fashion, non-blinded, through a sealed envelop randomization system.

Medical therapy withdrawal:

Medical therapy withdrawal will be conducted in 2 phases.

Phase 1:

This phase involves the withdrawal of the beta-blocker. The patient will be followed for signs of deterioration for a period of 6 months following the withdrawal.

Phase 2:

If there are no signs of deterioration the ACE/ARB inhibitor will be withdrawn as well. The patient will be followed up in 6 month for signs of deterioration. All other medical therapies other than beta-blocker and ACE inhibitors will continue until successful withdrawal of beta-blockers and ACE inhibitor is achieved.

Beta-blocker discontinuation:

The initial tapering off will occur over a 2week period. The beta -blocker will be discontinued by the end of the 2nd week.

For example: Metoprolol 100mg bid to Metoprolol 75mg bid for 5days. Followed by Metoprolol 50mg bid for 4 days, then Metoprolol 25 mg for 3 days and then completely discontinued.

ACE/ARB discontinuation:

The discontinuation of ACE/ARB will be similar to the beta-blockers. The doses will be tapered over a two-week period.

A supplementary chart of dose reduction is provided. The doses included are the standard medication doses.

Digoxin, diuretic, spironolactone will be discontinued if both the beta-blocker and ACE-ARB discontinuation has been well tolerated or if a clinical indication warrants the discontinuation. Up titration of therapies will not be permitted.

Additional therapy for SBP > 130 or DBP >80mmHg with non-ACE or beta blocker therapy will be considered.

Genotyping: Genetic analysis for DCM causing gene will be sent for the study patients. The genotyping is selective, patient will have the option to opt out the genetic analysis if they do not prefer having a genotyping done. All samples will be stored in a bio bank to maximum of 25 years. Two comparisons will be conducted on the genotyping:

1. The genetic typing for Patients with improved EF will be compared to the control group from the ongoing DCM cohort at the McGill University Health Center.
2. A second comparison between the patients within the withdrawal cohort. A comparison will be made between patients with rebound HF and the patient who did not HF with discontinuation of medical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with dilated cardiomyopathy (DCM) with an initial HFrEF < 40 % at presentation.
2. DCM with recovered LV function to > or = to 50% documented on 2 ECHO examinations, with the most recent ECHO examination within 1 year of enrolment.
3. Time from initial diagnosis of DCM more or equal to 24 month.
4. Last hospitalization for decompensated HF > 1year.

Exclusion criteria:

1. Ischemic cardiomyopathy
2. Other structural pathology such as: Hypertrophic cardiomyopathy, Valvular cardiomyopathy or congenital heart disease.
3. Last hospitalization for decompensated HF < 1year ago.
4. Previous sustained ventricle tachycardia or ventricle fibrillation (VF) arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Number of patients that become symptomatic | 1 year

SECONDARY OUTCOMES:
Number of patients that drop EF to <45% | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Giannetti, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta A, Goyal P, Bahl A. Frequency of recovery and relapse in patients with nonischemic dilated cardiomyopathy on guideline-directed medical therapy. Am J Cardiol. 2014 Sep 15;114(6):883-9. doi: 10.1016/j.amjcard.2014.06.021. Epub 2014 Jul 2. PMID 25084692
- [Background] Moon J, Ko YG, Chung N, Ha JW, Kang SM, Choi EY, Rim SJ. Recovery and recurrence of left ventricular systolic dysfunction in patients with idiopathic dilated cardiomyopathy. Can J Cardiol. 2009 May;25(5):e147-50. doi: 10.1016/s0828-282x(09)70497-0. PMID 19417864
- [Background] Zhang Y, Guallar E, Blasco-Colmenares E, Butcher B, Norgard S, Nauffal V, Marine JE, Eldadah Z, Dickfeld T, Ellenbogen KA, Tomaselli GF, Cheng A. Changes in Follow-Up Left Ventricular Ejection Fraction Associated With Outcomes in Primary Prevention Implantable Cardioverter-Defibrillator and Cardiac Resynchronization Therapy Device Recipients. J Am Coll Cardiol. 2015 Aug 4;66(5):524-31. doi: 10.1016/j.jacc.2015.05.057. PMID 26227190
- [Background] Blechman I, Arad M, Nussbaum T, Goldenberg I, Freimark D. Predictors and outcome of sustained improvement in left ventricular function in dilated cardiomyopathy. Clin Cardiol. 2014 Nov;37(11):687-92. doi: 10.1002/clc.22331. Epub 2014 Sep 18. PMID 25236761
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Basuray A, French B, Ky B, Vorovich E, Olt C, Sweitzer NK, Cappola TP, Fang JC. Heart failure with recovered ejection fraction: clinical description, biomarkers, and outcomes. Circulation. 2014 Jun 10;129(23):2380-7. doi: 10.1161/CIRCULATIONAHA.113.006855. Epub 2014 May 5. PMID 24799515
- [Background] Amos AM, Jaber WA, Russell SD. Improved outcomes in peripartum cardiomyopathy with contemporary. Am Heart J. 2006 Sep;152(3):509-13. doi: 10.1016/j.ahj.2006.02.008. PMID 16923422
- [Background] Waagstein F, Caidahl K, Wallentin I, Bergh CH, Hjalmarson A. Long-term beta-blockade in dilated cardiomyopathy. Effects of short- and long-term metoprolol treatment followed by withdrawal and readministration of metoprolol. Circulation. 1989 Sep;80(3):551-63. doi: 10.1161/01.cir.80.3.551. PMID 2548768
- [Background] Morimoto S, Shimizu K, Yamada K, Hiramitsu S, Hishida H. Can beta-blocker therapy be withdrawn from patients with dilated cardiomyopathy? Am Heart J. 1999 Sep;138(3 Pt 1):456-9. doi: 10.1016/s0002-8703(99)70147-x. PMID 10467195
- [Background] Hopper I, Samuel R, Hayward C, Tonkin A, Krum H. Can medications be safely withdrawn in patients with stable chronic heart failure? systematic review and meta-analysis. J Card Fail. 2014 Jul;20(7):522-32. doi: 10.1016/j.cardfail.2014.04.013. Epub 2014 Apr 18. PMID 24747201
- [Background] Pflugfelder PW, Baird MG, Tonkon MJ, DiBianco R, Pitt B. Clinical consequences of angiotensin-converting enzyme inhibitor withdrawal in chronic heart failure: a double-blind, placebo-controlled study of quinapril. The Quinapril Heart Failure Trial Investigators. J Am Coll Cardiol. 1993 Nov 15;22(6):1557-63. doi: 10.1016/0735-1097(93)90578-o. PMID 8227822
- [Background] Nicholls MG, Ikram H, Espiner EA, Maslowski AH, Scandrett MS, Penman T. Hemodynamic and hormonal responses during captopril therapy for heart failure: acute, chronic and withdrawal studies. Am J Cardiol. 1982 Apr 21;49(6):1497-501. doi: 10.1016/0002-9149(82)90367-8. PMID 6803564
- [Background] Konstam MA, Rousseau MF, Kronenberg MW, Udelson JE, Melin J, Stewart D, Dolan N, Edens TR, Ahn S, Kinan D, et al. Effects of the angiotensin converting enzyme inhibitor enalapril on the long-term progression of left ventricular dysfunction in patients with heart failure. SOLVD Investigators. Circulation. 1992 Aug;86(2):431-8. doi: 10.1161/01.cir.86.2.431. PMID 1638712
- [Background] Shammas NW, Harris ML, McKinney D, Hauber WJ. Digoxin withdrawal in patients with dilated cardiomyopathy following normalization of ejection fraction with beta blockers. Clin Cardiol. 2001 Dec;24(12):786-7. doi: 10.1002/clc.4960241207. PMID 11768743
- [Background] Khand AU, Rankin AC, Martin W, Taylor J, Gemmell I, Cleland JG. Carvedilol alone or in combination with digoxin for the management of atrial fibrillation in patients with heart failure? J Am Coll Cardiol. 2003 Dec 3;42(11):1944-51. doi: 10.1016/j.jacc.2003.07.020. PMID 14662257
- [Background] Cuenca S, Ruiz-Cano MJ, Gimeno-Blanes JR, Jurado A, Salas C, Gomez-Diaz I, Padron-Barthe L, Grillo JJ, Vilches C, Segovia J, Pascual-Figal D, Lara-Pezzi E, Monserrat L, Alonso-Pulpon L, Garcia-Pavia P; Inherited Cardiac Diseases Program of the Spanish Cardiovascular Research Network (Red Investigacion Cardiovascular). Genetic basis of familial dilated cardiomyopathy patients undergoing heart transplantation. J Heart Lung Transplant. 2016 May;35(5):625-35. doi: 10.1016/j.healun.2015.12.014. Epub 2016 Jan 6. PMID 26899768
- [Background] Sheppard R, Hsich E, Damp J, Elkayam U, Kealey A, Ramani G, Zucker M, Alexis JD, Horne BD, Hanley-Yanez K, Pisarcik J, Halder I, Fett JD, McNamara DM; IPAC Investigators. GNB3 C825T Polymorphism and Myocardial Recovery in Peripartum Cardiomyopathy: Results of the Multicenter Investigations of Pregnancy-Associated Cardiomyopathy Study. Circ Heart Fail. 2016 Mar;9(3):e002683. doi: 10.1161/CIRCHEARTFAILURE.115.002683. PMID 26915373
- [Background] Ware JS, Li J, Mazaika E, Yasso CM, DeSouza T, Cappola TP, Tsai EJ, Hilfiker-Kleiner D, Kamiya CA, Mazzarotto F, Cook SA, Halder I, Prasad SK, Pisarcik J, Hanley-Yanez K, Alharethi R, Damp J, Hsich E, Elkayam U, Sheppard R, Kealey A, Alexis J, Ramani G, Safirstein J, Boehmer J, Pauly DF, Wittstein IS, Thohan V, Zucker MJ, Liu P, Gorcsan J 3rd, McNamara DM, Seidman CE, Seidman JG, Arany Z; IMAC-2 and IPAC Investigators. Shared Genetic Predisposition in Peripartum and Dilated Cardiomyopathies. N Engl J Med. 2016 Jan 21;374(3):233-41. doi: 10.1056/NEJMoa1505517. Epub 2016 Jan 6. PMID 26735901